CLINICAL TRIAL: NCT03576092
Title: Lung Ultrasound Patterns in Late Third-trimester Gravidas With and Without Preeclampsia
Brief Title: Lung Ultrasound Patterns Preeclampsia
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: HS16-0447
Record Dates: First submitted 2018-05-29; First posted 2018-07-03 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Pregnancy Complications; Ultrasound Therapy; Complications; Pulmonary Disease; Pulmonary Edema
MeSH Terms: conditions — Pregnancy Complications; Lung Diseases; Pulmonary Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Pregnancy: Healthy gestational age-matched pregnant patients from 32 - 41 weeks without a diagnosis of preeclampsia.
  Interventions: Diagnostic Test: Lung Ultrasound
- Preeclampsia Pregnancy: Pregnant patients from 32 - 41 weeks with a diagnosis of preeclampsia based on standard criteria as outlined by the American Congress of Obstetrics and Gynecology (ACOG).
  Interventions: Diagnostic Test: Lung Ultrasound

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound — Lung sonography will be performed on a SonoSite portable ultrasound machine with a C60e 5 - 2 MHx 30cm probe using a modified standard technique examining four lung regions; anterior mid-clavicular high and low on left and right sides, and one on each side posteriorly) in the semi-recumbent position.

SUMMARY:
Evaluation of lung ultrasound as a diagnostic tool in pregnant patients.

DETAILED DESCRIPTION:
The objective of this study is to evaluate lung ultrasound as a tool in pregnant patients. This tool has not been well studied in pregnancy but has the potential to detect pulmonary edema in patients with preeclampsia before they become critically ill. In addition, the presence of pulmonary edema is a criterion for the diagnosis for severe preeclampsia, and if detected early, may change management and decrease morbidity in these patients. The investigators hypothesize that healthy pregnant women and women with preeclampsia in the third trimester have normal lung ultrasound patterns in the absence of clinical signs or symptoms of poor lung aeration.

The investigators propose a prospective cross-sectional study to compare pregnant patients with and without a diagnosis of preeclampsia treated at the Long Island Jewish Medical Center (LIJ) and North Shore University Hospital (NSUH) from August 2016 - May 2018. A cohort of healthy gestational age-matched pregnant patients from 32 - 41 weeks without a diagnosis of preeclampsia will serve as controls. Inclusion criteria include singleton pregnancies over 31 6/7 weeks gestational age treated at LIJ or NSUH. Exclusion criteria include age less than 18 years and refusal to participate in the study. Informed consent will be obtained for all study participants.

A diagnosis of preeclampsia will be made based on standard criteria as outlined by the American Congress of Obstetrics and Gynecology (ACOG). Interstitial edema will be defined as an ultrasound finding of three or more B-lines in an interstitial space in two or more lung regions. B-line dominant lung fields are suggestive of alveolar interstitial syndrome. The clinical diagnosis of pulmonary edema is based on findings including dyspnea, tachypnea, tachycardia, hypoxemia (measured by non-invasive pulse oximeter), and diffuse crackles on lung exam. The patient characteristics and ultrasound findings will be compared between the cohort of preeclamptic patients and healthy controls. A secondary analysis will be performed on the images that were obtained before and after magnesium sulfate therapy in patients diagnosed with preeclampsia with severe features to determine the effect on sonographic findings. If a preeclamptic patient received a chest x-ray as part of her management plan because of a clinical suspicion of pulmonary edema, the reported results will be collected and compared to lung sonogram results.

Lung sonography will be performed on a SonoSite portable ultrasound machine with a C60e 5 - 2 MHx 30cm probe using a modified standard technique examining four lung regions; anterior mid-clavicular high and low on left and right sides, and one on each side posteriorly) in the semi-recumbent position. Still images and video clips will be reviewed by an expert in lung ultrasound who is blinded to the patients' clinical information (Dr. Seth Koenig). Lung sonography will be performed on two occasions for each preeclamptic patient who is treated with magnesium sulfate; 1) at the time of diagnosis of preeclampsia, and 2) after completion of magnesium sulfate bolus. Lung sonography will be performed on only one occasion for gestational age-matched controls and for preeclamptic patients who are not treated with magnesium sulfate. Patients will not be given a diagnosis of pulmonary edema nor will their management plans be altered based on the results of the lung sonography performed for this study.

Data will be collected and stored in RedCap. The investigators will collect data on patient demographics, past medical and surgical history, blood pressure measurements at time of diagnosis, results of routine lab values that are drawn for evaluation of preeclamptic patients, and the review of four ultrasound examination regions to determine if they are B-line dominant or A-line dominant. Descriptive statistics and appropriate comparison tests will be used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Singleton pregnancy
* 32 0/7 weeks - 41 6/7 weeks gestational age

Exclusion Criteria:

* Inability to provide informed consent
* Refusal to participate
* Already treated for acute lung pathology prior to enrollment
* Cognitive impairment that precluded understanding of research procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject population is 262 pregnant female participants between ages 18 to approximately 49 years old. Pregnant patients must be used in the study population because the objective is to evaluate lung ultrasound as a tool in the pregnant population.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-05-20 (Actual)

PRIMARY OUTCOMES:
Positive Lung Ultrasound Study | At time of lung ultrasound study, through study completion from August 2016 - May 2018.
  ultrasound finding of three or more B-lines in an interstitial space in two or more lung regions.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco PA, Cianciulli TF. Pulmonary Edema Assessed by Ultrasound: Impact in Cardiology and Intensive Care Practice. Echocardiography. 2016 May;33(5):778-87. doi: 10.1111/echo.13182. Epub 2016 Feb 3. PMID 26841270
- [Background] Pachtman S, Koenig S, Meirowitz N. Detecting Pulmonary Edema in Obstetric Patients Through Point-of-Care Lung Ultrasonography. Obstet Gynecol. 2017 Mar;129(3):525-529. doi: 10.1097/AOG.0000000000001909. PMID 28178063
- [Background] Dennis AT, Solnordal CB. Acute pulmonary oedema in pregnant women. Anaesthesia. 2012 Jun;67(6):646-59. doi: 10.1111/j.1365-2044.2012.07055.x. Epub 2012 Mar 15. PMID 22420683
- [Background] Inchingolo R, Smargiassi A, Mormile F, Marra R, De Carolis S, Lanzone A, Valente S, Corbo GM. Look at the lung: can chest ultrasonography be useful in pregnancy? Multidiscip Respir Med. 2014 Jun 6;9(1):32. doi: 10.1186/2049-6958-9-32. eCollection 2014. PMID 24936303
- [Background] Malek G, Drygalska A, Kober J, Wawrzynska L, Debski R, Dabrowski M, Torbicki A. [Chest ultrasound in the diagnosis of pulmonary embolism in a pregnant patient - a case report]. Pneumonol Alergol Pol. 2009;77(6):560-4. Polish. PMID 20013708
- [Background] Samol JM, Lambers DS. Magnesium sulfate tocolysis and pulmonary edema: the drug or the vehicle? Am J Obstet Gynecol. 2005 May;192(5):1430-2. doi: 10.1016/j.ajog.2005.02.093. PMID 15902128
- [Background] Sibai BM, Mabie BC, Harvey CJ, Gonzalez AR. Pulmonary edema in severe preeclampsia-eclampsia: analysis of thirty-seven consecutive cases. Am J Obstet Gynecol. 1987 May;156(5):1174-9. doi: 10.1016/0002-9378(87)90135-9. PMID 3578433
- [Background] Volpicelli G, Mussa A, Garofalo G, Cardinale L, Casoli G, Perotto F, Fava C, Frascisco M. Bedside lung ultrasound in the assessment of alveolar-interstitial syndrome. Am J Emerg Med. 2006 Oct;24(6):689-96. doi: 10.1016/j.ajem.2006.02.013. PMID 16984837